CLINICAL TRIAL: NCT03126422
Title: Effects of Different Doses of Dexmedetomidine on Fentanyl-induced Cough
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yangzhou University (Other)
Responsible Party: Principal Investigator, Zhuan Zhang, Director, Yangzhou University
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 20170413
Record Dates: First submitted 2017-04-14; First posted 2017-04-24 (Actual); Last update posted 2017-07-05 (Actual); Status verified 2017-07

CONDITIONS: Fentanyl-induced Cough
MeSH Terms: interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Dexmedetomidine 0 μg/kg/min (Experimental)
  Interventions: Drug: Dexmedetomidine
- Dexmedetomidine 0.03 μg/kg/min (Experimental)
  Interventions: Drug: Dexmedetomidine
- Dexmedetomidine 0.06 μg/kg/min (Experimental)
  Interventions: Drug: Dexmedetomidine
- Dexmedetomidine 0.09 μg/kg/min (Experimental)
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine — Pretreatment of different doses of dexmedetomidine

SUMMARY:
The investigators aimed to investigate the effects of pretreatment with different doses of dexmedetomidine on the cough caused by fentanyl during anesthetic induction.

Patients undergoing elective surgeries under general anesthesia will be randomly allocated to 4 groups (n = 60, each group). Dexmedetomidine 0, 0.03, 0.06, and 0.09 μg/kg/min will be pump-administered in 10 mins to groups I, II, III, and IV, respectively, followed by the induction of general anesthesia with intravenous fentanyl 4 μg/kg. The incidences and severity of cough that occurred within 2 min after the injection of fentanyl will be recorded, and the incidences of cardiovascular adverse events that occurred between the administration of the dexmedetomidine infusion and 2 min after tracheal intubation will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective surgeries under general anesthesia.

Exclusion Criteria:

* Patients with contraindications of dexmedetomidine.
* Patients younger than 18 years old and older than 65 years old.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2017-05-01 (Actual); Primary Completion 2017-09-01 (Estimated); Study Completion 2017-09-01 (Estimated)

PRIMARY OUTCOMES:
The incidence of cough | After the infusion of dexmedetomidine up to 10 minutes
  Yes or No
The time of cough | After the infusion of dexmedetomidine up to 10 minutes
  After the infusion of dexmedetomidine up to 10 minutes
The severity of cough | After the infusion of dexmedetomidine up to 10 minutes
  minor, moderate, severe
The occurence of adverse effects of dexmedetomidine | After the infusion of dexmedetomidine up to 10 minutes
  bradycardia, hypotension, hypertension

CONTACTS AND LOCATIONS:
Locations (1):
- the Affiliated Hospital of Yangzhou University, Yangzhou University, Yangzhou, Jiangsu, China

REFERENCES:
- [Derived] Zhou W, Zhang D, Tian S, Yang Y, Xing Z, Ma R, Zhou T, Bao T, Sun J, Zhang Z. Optimal dose of pretreated-dexmedetomidine in fentanyl-induced cough suppression: a prospective randomized controlled trial. BMC Anesthesiol. 2019 Jun 1;19(1):89. doi: 10.1186/s12871-019-0765-z. PMID 31153360